CLINICAL TRIAL: NCT06940752
Title: VINTAGE (Ventricular Intramyocardial Navigation for Tachycardia Ablation Guided by Electrograms) Using Commercial Off-The-Shelf (COTS) Catheters, Early Feasibility Study
Brief Title: VINTAGE (Ventricular Intramyocardial Navigation for Tachycardia Ablation Guided by Electrograms) Using Commercial Off-The-Shelf (COTS) Catheters
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 10002320; 002320-H
Record Dates: First submitted 2025-04-22; First posted 2025-04-23 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12-09

CONDITIONS: Ventricular Arrhythmia
Keywords: ablation therapy; CATHETERIZATION

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- VINTAGE Arm (Experimental): Non-surgical catheter approach called VINTAGE will be used to treat ventricular arrhythmias arising from difficult-to-reach portions of the heart.
  Interventions: Device: VINTAGE (Ventricular Intramyocardial Navigation for Tachycardia Ablation Guided by Electrograms)

INTERVENTIONS:
Device: VINTAGE (Ventricular Intramyocardial Navigation for Tachycardia Ablation Guided by Electrograms) — Non-surgical catheter approach called VINTAGE will be used to treat ventricular arrhythmias arising from difficult-to-reach portions of the heart.

SUMMARY:
Background:

Ventricular arrhythmia is an abnormal pulse rhythm that starts in the lower part of the heart (ventricles). Treatment includes ablation; ablation uses heat to destroy small portions of the heart that are causing short circuits in the normal heartbeats. But ablation does not always work well because some parts of the heart are hard to reach with current tools. Researchers want to try a new method called VINTAGE (ventricular intramyocardial navigation for tachycardia ablation guided by electrograms). VINTAGE may be better able to treat portions of the heart that are harder to reach with standard techniques.

Objective:

To test VINTAGE in people with ventricular arrhythmia.

Eligibility:

People aged 21 years and older with ventricular arrhythmia that did not respond to standard treatment.

Design:

Participants will have baseline tests. They will have blood tests and tests of their heart function. They will have imaging scans. They will complete a health questionnaire.

Participants will undergo the VINTAGE procedure. They will be either completely or partially asleep. Doctors will insert tubes through large blood vessels in the groin. Tubes may also be inserted through the chest and wrist. They will use x-rays and ultrasound to guide tubes and guidewires directly into the heart muscle to do the ablation.

Participants will stay in the hospital 1 or more nights after the procedure.

Participants will have 3 follow-up visits over 6 months. These visits are for standard care after heart ablation. They will include blood tests, imaging scans, and tests of heart function. Participants may also wear a device to monitor their heart rhythms at home.

DETAILED DESCRIPTION:
Ventricular arrhythmias cause heart damage or death. Ventricular arrhythmias usually arise from small zones of the heart that contribute a short circuit or errant stimulus. Ventricular arrhythmias may be reduced or abolished by non-surgical catheter procedures to heat and destroy the small portions of the heart that contribute a short circuit or abnormal pacemaker. However, not all portions of the heart can physically be reached for catheter treatment.

We have developed a new non-surgical catheter approach called VINTAGE (Ventricular Intramyocardial Navigation for Tachycardia Ablation Guided by Electrograms) to treat ventricular arrhythmias arising from difficult-to-reach portions of the heart. In VINTAGE, catheter tools are moved inside the walls of the beating heart to reach treatment targets. In a small number of patients who failed prior catheter treatment of ventricular arrhythmia, VINTAGE effectively suppressed the ventricular arrhythmia or abnormal pacemaker in most.

The purpose of this research protocol is to test VINTAGE more carefully in people with ventricular arrhythmias who have failed prior catheter ablation. In this protocol, we will use catheter tools that are commercially available but are not designed or approved for use in VINTAGE.

ELIGIBILITY:
* INCLUSION CRITERIA:

Candidates must meet all of the following criteria:

* Age >= 21 years
* Undergoing planned repeat radiofrequency catheter ablation for ventricular arrhythmias (Having failed a previous attempt at catheter ablation and at least one antiarrhythmic drug for ventricular arrhythmias)
* Ventricular arrhythmia COHORT 1:

  * Monomorphic ventricular tachycardia
  * Has an implanted cardioverter defibrillator (ICD)
  * Hospital admission for ventricular tachycardia since most recent ablation attempt
* Ventricular arrhythmia COHORT 2:

  --Monomorphic (unifocal), frequent, premature ventricular contraction, >=15% burden
* Naive pericardium (no prior cardiac surgery)
* Either of

  * Symptomatic (intolerable palpitation, syncope, fatigue, dyspnea, heart failure, hospital admission for ventricular arrhythmia, appropriate ICD discharge, appropriate antitachycardia pacing), OR
  * Left ventricular ejection fraction < 0.50
* Willing to return for all scheduled follow-up activities, and eligible or able to undergo required protocol and testing

EXCLUSION CRITERIA:

* Does not consent to participate, or unable to consent to participate
* Left ventricular ejection fraction < 0.20
* Hemodynamic instability or emergency procedure
* Requires planned temporary mechanical circulatory device (such as percutaneous left ventricular assist device or intraaortic balloon counterpulsation pump)
* Pregnant
* eGFR < 30 mL/min/1.73m^2 or end-stage renal failure requiring renal replacement therapy
* Survival despite successful procedure expected < 6 mo

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
VT COHORT: Freedom from appropriate implanted cardioverter-defibrillator (ICD) shocks or hospital admission due to recurrent VT | 6 months
  The primary endpoint for VT Cohort is freedom from appropriate implanted cardioverter-defibrillator (ICD) shocks or hospital admission due to recurrent VT at 6 months.
PVC COHORT: Reduction in PVC burden | 6 months
  The primary endpoint for participants treated for PVC Cohort is reduction in PVC burden at 6 months.

SECONDARY OUTCOMES:
Freedom from major adverse cardiovascular events | Time of discharge
  The secondary endpoint is freedom from major adverse cardiovascular events at the time of discharge from the index VINTAGE procedure. This excludes VINTAGE-related pericarditis and pericardial effusion not requiring secondary intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Lederman, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD that underline results in a publication will be shared. Medical images will not be shared because of intrinsic inability to protect confidentiality with reasonable effort.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available by the end of the project or protocol or at the time of associated publication.
Access Criteria: BioData Catalyst is supported by NHLBI and access to data is controlled by the NHLBI Data Access Committee (DAC) utilizing the database of Genotypes and Phenotypes (dbGaP) permissions infrastructure. In order to access controlled-access data in BioData Catalyst, an investigator must have an approved Data Access Request (DAR) in dbGaP.